CLINICAL TRIAL: NCT04373603
Title: Randomized Controlled Trial Evaluating the Co-Administration of HA and TXA in Facial Filler
Brief Title: Use of Tranexamic Acid in Facial Fillers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed prior to opening to enrollment, due to funding availability for study
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-0573; A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison); Protocol version 0.11 (Other: HS-IRB UW, Madison)
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Injection Site Bruising
Keywords: patient satisfaction; plastic surgery
MeSH Terms: conditions — Patient Satisfaction | interventions — Tranexamic Acid; Sodium Chloride; Hyaluronic Acid; Hyaluronoglucosaminidase

STUDY DESIGN:
Intervention Model Description: half face study where participant serves as own control, intervention on one side of the face, control on the other
Who Masked: Participant, Investigator
Masking Description: side of face for treatment is randomized and double blinded to the participant and physician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: HA plus TXA (Experimental): HA will be diluted with TXA using a Leur-Lok hub in a ratio of 1.0 mL HA filler to 0.2 mL TXA (100mg/mL)
  Interventions: Drug: Tranexamic acid; Drug: Hyaluronic acid
- Control: HA plus Saline (Placebo Comparator): HA will be diluted with saline in a ratio of 1.0 mL HA filler to 0.2 mL saline
  Interventions: Other: Saline; Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Tranexamic acid — TXA is a synthetic lysine analogue that inhibits the activation of plasminogen to plasmin, thus inhibiting degradation of fibrin clots and serving as an antifibrinolytic
  Other Names: TXA
  Arms: Intervention: HA plus TXA
Other: Saline — sodium chloride and water for use as control
  Arms: Control: HA plus Saline
Drug: Hyaluronic acid — Hyaluronidase is a spreading or diffusing substance which modifies the permeability of connective tissue through the hydrolysis of hyaluronic acid, a polysaccharide found in the intercellular ground substance of connective tissue
  Other Names: HA; Hyaluronidase

SUMMARY:
The overall purpose of this study is to evaluate the safety and efficacy of co-administration of tranexamic acid (TXA) with hyaluronic acid (HA) in reducing swelling, bruising and pain after facial injection. This will be done by comparing HA to HA+TXA in participants undergoing facial filler injections. Patients undergoing facial filler injections almost always have the same type of injection performed bilaterally in order to maintain symmetry. This provides a unique opportunity where participants can serve as their own controls. Participants will be injected with HA on half of their face and the other half of the face will be injected with HA+TXA. Swelling, bruising, pain, and overall satisfaction will be assessed using participant self-reported surveys, physician surveys, and review of medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 but less than or equal to 89 years.
* Medically appropriate to undergo elective facial filler injection at UW Health by principal investigator
* English speaking

Exclusion Criteria:

* Minors or under the age of 18
* Patient over the age of 89
* Pregnant or breast-feeding women
* Individuals unable to give consent due to another condition such as impaired decision-making capacity.
* Participants with a history of a thrombotic event (DVT, PE, stroke, MI) or genetic disorder that increases risk of thrombosis
* Concurrent use of estrogen
* Participant undergoing unilateral facial filler injections
* Participants with history of hypersensitivity to TXA or any of the other ingredients
* Participants that are on current therapeutic anticoagulation therapy
* Participants with stage 2 or greater renal failure
* Participants on hemo- or peritoneal dialysis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Intensity of Bruising Score | Post procedure day 7
  Participant reported intensity of bruising score on a 5 point Likert scale where 1 is no bruising and 5 is severe bruising.

SECONDARY OUTCOMES:
Intensity of Bruising Score | Post procedure day 1
  Participant reported intensity of bruising score on a 5 point Likert scale where 1 is no bruising and 5 is severe bruising.
Intensity of Bruising Score | Post procedure day 30
  Participant reported intensity of bruising score on a 5 point Likert scale where 1 is no bruising and 5 is severe bruising.
Intensity of Swelling Score | Post procedure day 1
  Participant reported intensity of swelling score on a 5 point Likert scale where 1 is no swelling and 5 is severe swelling.
Intensity of Swelling Score | Post procedure day 7
  Participant reported intensity of swelling score on a 5 point Likert scale where 1 is no swelling and 5 is severe swelling.
Intensity of Swelling Score | Post procedure day 30
  Participant reported intensity of swelling score on a 5 point Likert scale where 1 is no swelling and 5 is severe swelling.
Pain Score | Post procedure day 1
  Participants will rate their pain on a scale of 0-10 where 0 is no pain and 10 is the highest pain.
Pain Score | Post procedure day 7
  Participants will rate their pain on a scale of 0-10 where 0 is no pain and 10 is the highest pain.
Pain Score | Post procedure day 30
  Participants will rate their pain on a scale of 0-10 where 0 is no pain and 10 is the highest pain.
Participant Satisfaction Score | Post procedure day 1
  Participants will rate their satisfaction on a 5 point Likert scale where 1 is completely dissatisfied and 5 is completely satisfied.
Participant Satisfaction Score | Post procedure day 7
  Participants will rate their satisfaction on a 5 point Likert scale where 1 is completely dissatisfied and 5 is completely satisfied.
Participant Satisfaction Score | Post procedure day 30
  Participants will rate their satisfaction on a 5 point Likert scale where 1 is completely dissatisfied and 5 is completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Afifi, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No